CLINICAL TRIAL: NCT02373501
Title: Extra - Abdominal Versus Intra - Abdominal Repair of the Uterine Incision at Cesarean Section
Acronym: EKAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Elias Castel, Senior Resident Obstetrics and Gynocology, Dr. Elias Castel, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-13-0494-EC-CTIL
Record Dates: First submitted 2013-07-29; First posted 2015-02-27 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Cesarean Wound Repair
Keywords: caesarean delivery; uterine incision repair

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intra-abdominal repair (Experimental): intra-abdominal repair of uterine incision, after delivery of the fetus and the placenta.
  Interventions: Procedure: Intra-abdominal repair
- extra-abdominal repair (Experimental): extra-abdominal repair of uterine incision, after delivery of the fetus and the placenta.
  Interventions: Procedure: Extra-abdominal repair

INTERVENTIONS:
Procedure: Intra-abdominal repair — Intra abdominal repair of uterine incision
  Arms: intra-abdominal repair
Procedure: Extra-abdominal repair — Extra abdominal repair of uterine incision
  Arms: extra-abdominal repair

SUMMARY:
To evaluate the effects of extra-abdominal repair of the uterine incision compared to intra-abdominal repair, and to study is there superiority of one technique over the other in terms of primary outcomes - operative( up to 4 hours after beginning of anesthesia) and post operative ( until day 4 after operation ) measurements , secondary outcomes, long-term outcomes and subjective outcomes.

PRIMARY OUTCOMES:

Intra - operative ( during the operation up to 4 hours from anesthesia )

* nausea and vomiting
* intraoperative hypotension
* intraoperative pain

Post operative ( 4 hours from anesthesia and until release from hospital )

* Blood transfusion
* Venous thromboembolism
* Febrile Morbidity
* Endometritis
* Wound Infection
* Death

Subjective measures:

* complain of pain 1-10 on day 1 post operative
* time until walking
* number of Days until having bowel movement
* overall satisfactory

SECONDARY OUTCOMES:

* Operative time
* Estimated blood loss ( ebl ) - hemoglobin levels
* Hospital stay

DETAILED DESCRIPTION:
Cesarean section (CS) delivery is one of the most frequent surgical procedures to be performed worldwide and rates of CS delivery are increasing. In the late 80's, the rate of caesarean deliveries was 10-13 % in most of the big hospitals in Israel, and today it reaches up to 20-25% of all deliveries.

Numerous different surgical techniques for caesarean section delivery have been described, and the debate about the optimal caesarean technique to minimize surgical morbidity is ongoing.

One of the more controversial issues regarding caesarean technique is the manner by which uterine repair is conducted after delivery of the infant(s) and placenta.

Two techniques are being used depending on the uterus position during repairmen : In situ within the peritoneal cavity (intra- abdominal repair) or temporarily exteriorized onto the mother's abdomen (extra- abdominal repair).

Arguments in favor of temporary exteriorization include better visualization of any uterine extensions and more rapid uterine repair with consequent reductions in both operative time and intraoperative blood loss. Opponents of extraabdominal repair argue that this technique increases rates of intraoperative nausea and vomiting, adnexal trauma on replacement, possible infection, and venous air embolism (VAE) .

On this study the investigators prospectively recruit women who are about to be electively operated. The patients will be randomized into two groups - extra- abdominal versus intra-abdominal uterine repair using computer randomization. Different charts will be for first CS delivery versus recurrent CS delivery. The patient won't know to which group she was designated . On day three after operation - she will be asked to fill out questionnaire with one of the investigators for subjective measurements

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* term pregnancy

Exclusion Criteria:

* chorioamnionitis
* uterine rupture
* hysterotomy - adhesiolysis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
nausea and vomiting | during operation- 4 hours from anasthesia
intraoperative hypotension | during operation- 4 hours from anasthesia
intraoperative pain | during operation- 4 hours from anasthesia
Blood transfusion | during operation- 4 hours from anasthesia
Venous thromboembolism | durind operation - 4 hours from anasthesia
Febrile Morbidity | post operative - untill release from hospitalization usually day 4
Endometritis | post operative- untill release from hospitalization usually day 4
Wound Infection | post operative- untill release from hospitalization usually day 4
Death | post operative - untill release from hospitalization usually day 4

SECONDARY OUTCOMES:
Operative time | operative time - since anasthesia untill closure of skin
Estimated blood loss ( ebl ) - HGB levels | operative- 4 hours from anasthesia
Hospital stay | post operative

OTHER OUTCOMES:
complain of pain 1-10 on day 1 post operative | post operative - on day 3 post operative
time from surgery until first walking | post operative - during hospitalization
number of Days until having bowel movement, | post operative - during hospitalization
overall satisfactory | post operative - during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Elias Castel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Jacob CE, Pasquier JC. Extraabdominal vs intraabdominal uterine repair at cesarean delivery: a metaanalysis. Am J Obstet Gynecol. 2010 Apr;202(4):e10-1; author reply e11. doi: 10.1016/j.ajog.2009.10.879. Epub 2009 Dec 22. No abstract available. PMID 20022585